CLINICAL TRIAL: NCT05454046
Title: Food & Fertility - Does Food Intake Affect Your Fertility?
Brief Title: Food Intake Among Women and Men in Fertility Treatment
Acronym: Food&Fertility
Status: Recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Statens Serum Institut (Other); Herlev and Gentofte Hospital (Other); Regional Hospital Skive (Unknown); Regionshospitalet Horsens (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Ulrik Schiøler Kesmodel, Professor, Aalborg University Hospital
Other Study IDs: AGR-2019-731-9666
Record Dates: First submitted 2022-07-08; First posted 2022-07-12 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Infertility
Keywords: Fertility; Assisted reproductive techniques; Food; Diet; Dietary supplements; Semen quality; Live birth
MeSH Terms: conditions — Infertility | interventions — Menogaril

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women
  Interventions: Other: Food intake among women and men in fertility treatment
- Men
  Interventions: Other: Food intake among women and men in fertility treatment

INTERVENTIONS:
Other: Food intake among women and men in fertility treatment — Filling in an FFQ

SUMMARY:
Worldwide infertility is highly prevalent and lifestyle factors, such as food intake, could have an essential role in the success of a fertility treatment. The literature is not consistent and adequate for recommendations to the increasing number of women and men of reproductive age who ask for lifestyle guidance. Therefore, the aims of the Food & Fertility study will be to investigate the association between food intake and semen quality, pregnancy- and live birth rates in women and men undergoing assisted reproductive technology (ART) treatment.

DETAILED DESCRIPTION:
The Food & Fertility study is a multicenter prospective cohort study which is planned to enroll a total of 4000 women and men between 2022 and 2024. The data collection will take place in four fertility clinics through a web-based food frequency questionnaire (FFQ). Data on sperm quality and pregnancy- and live birth rates will be obtained from medical records and national registers.

ELIGIBILITY:
Inclusion Criteria:

* Women and men undergoing fertility treatment: in vitro fertilization (IVF), intracytoplasmatic sperm injection (ICSI), frozen-thawed embryo transfer (FET) or intrauterine insemination (IUI).
* Availability of a semen sample analyzed 3 months before or after filling in the FFQ.
* Read and understands Danish.

Exclusion Criteria:

* Treatment with double donation (both semen and oocyte donation)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women and men undergoing ART treatment or intrauterine insemination (IUI) at the fertility clinics at Aalborg University Hospital, Herlev University Hospital, and at the Regional Hospitals in Horsens and Skive will be invited to participate in the study (n=4000).
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Probability of live birth | From filling out the FFQ to birth (approximately 9-10months)
Probability of pregnancy | From filling out the FFQ to end of treatment cycle (approximately 3 weeks)
Semen quality | +/- 3 months from filling out the FFQ

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Herlev Hospital Copenhagen, Herlev
  - Regional Hospital Horsens, Horsens
  - Odense University Hospital, Odense
  - Regional Hospital Skive, Skive

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buhl Borgstrom MB, Ahrendt Bjerregaard A, Olsen SF, Gabrielsen A, Humaidan P, Kesmodel US. Food & Fertility Study: study protocol for a Danish multicentre prospective cohort study investigating the association between food intake and semen quality, pregnancy and birth outcomes in infertile women and men. BMJ Open. 2023 Jul 4;13(7):e068354. doi: 10.1136/bmjopen-2022-068354. PMID 37407049